CLINICAL TRIAL: NCT06902194
Title: Mucosal Surveillance and Immunology of Respiratory Pathogens in South African Children Post the COVID-19 Pandemic
Brief Title: To Evaluate Mucosal and Systematic Immune Response to Acute Respiratory Tract Infections of South African Children
Acronym: Muco-Kids
Status: Recruiting | Type: Observational
Sponsor: Desmond Tutu TB Centre (Other)
Collaborators: European Union (Other)
Responsible Party: Sponsor
Other Study IDs: N24/08/097-ID31271; VERDI (101045989) (Other Grant/Funding Number: Europe Horizon 2020, European Union)
Record Dates: First submitted 2025-02-03; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-02

CONDITIONS: Respiratory Tract Infections (RTI); Mucosal Immunity
Keywords: Mucosal immunity; Mucosal immunology; Respiratory tract infections; Saliva
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and paxgene samples, as well as saliva and nasopharyngeal aspirate specimens will be collected and stored.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Acute RTIs: Children aged 0-13 years presenting with acute respiratory tract infections to Tygerberg Hospital.

SUMMARY:
The goal of this observational study is to answer a few questions about respiratory tract infections in South African children:

1. How do children with COVID-19 and other respiratory (chest, throat, ear or nose) germs show symptoms? What signs should be looked for, and which children are more likely to get seriously ill? Are there any new germs that haven't been discovered yet? Can immune cells in saliva predict which children will get more severe disease?
2. The body's immune response (soldier- cells) in blood and saliva (spit) will be studied.
3. What is the short-term effect of COVID-19 and other respiratory viruses/ germs on the breathing (lung function) of children?
4. What is the impact of respiratory germs on the quality of life in children and their families? The investigators aim to recruit a minimum of 250 children with respiratory pathogens.

DETAILED DESCRIPTION:
This observational cohort study will include children aged 0-13 years with acute respiratory tract infections who present to Tygerberg Hospital (TBH) for routine care. Key routine care data, including vaccination history, detailed medical history, and treatments received during hospital admission (such as oxygen therapy, antiviral medication, antibiotics, or other supportive drugs), will be documented in case report forms (CRFs).

South Africa has a high burden of tuberculosis and HIV infection, and it is important to study respiratory tract infections in this population.

Children aged 0-13 years will be recruited from Tygerberg Hospital (TBH), which functions as a regional referral center for the surrounding health sub-districts, including Northern, Tygerberg, Khayelitsha, and Eastern, collectively serving over 30% of the metropolitan population (3.5 million residents). Additionally, TBH acts as a tertiary-level referral center for paediatric emergencies, infectious diseases, and pulmonology.

Children with acute respiratory symptoms who present to TBH will be enroled in the study, provided they have been hospitalised for less than 72 hours, consent has been obtained from both the caregiver and child (where applicable), and there are no medical contraindications to collecting respiratory samples.

This study will be implemented within routine care services and clinical and laboratory data collected for routine care will be used for research. The research team will collect additional data and samples.

Additional samples collected at enrolment will include blood, mucus, and saliva. Additional saliva samples will be taken on the second and third days of hospital admission, as well as at discharge.

About one and a half teaspoons of blood will be taken on enrolment to perform the following tests:

1. Antibody analysis

   1. Antibodies targeting common respiratory pathogens, as well as polyreactive (non-specific) antibodies
   2. Total IgM/IgG/IgA
2. PAXgene for transcriptomics. Transcriptomics is the study of all the RNA molecules (called the transcriptome) in a cell, tissue, or organism at a given time. It helps scientists understand which genes are active (turned on) and how much they are being used.

Nasopharyngeal aspirates will be used to collect mucus. A thin tube will be inserted into one nostril to the back of the throat and the mucus will be sucked up into a tube.

Polymerase chain reaction (PCR) will be used to look for common respiratory viruses. Samples will also be saved for later metagenomic sequencing (looking for all the viruses, bacteria and fungi that are present in the sample).

Saliva will be collected at enrolment, on the second and third day of admission and at discharge, by leaving a cottonwool sample in the mouth until it is soaked. The antibodies in saliva will be compared to those in the blood. In addition, mucosal immune markers such as cytokines will be measured.

Baseline and follow-up questionnaires will collect detailed clinical information.

1. Standard symptomatology questionnaires

   1. Signs and symptoms of presenting illness will be recorded, including upper and lower respiratory tract symptoms and fever. Previous medical history of respiratory symptoms including recurring respiratory symptoms, chronic illnesses (including TB and HIV) and the use of chronic medication.
   2. Constitutional factors including gender, birth weight, gestational age at birth, HIV exposure status and family history of asthma or atopy.
   3. Environmental factors including TB exposure, tobacco smoke exposure during and after pregnancy, and indoor cooking.
   4. Nutritional status information regarding diet, and growth preceding hospitalisation as evidenced in the Road-To-Health Card.
   5. Microbiome-specific questions, birth history, diet.
2. Quality of life (QoL, standard measure by age cohort). Standardised health-related quality of life questionnaire

Statistical Analysis:

The investigators intend to enrol between 200-300 South African children (see power calculation below). This will allow the use of a targeted protein marker approach in combination with antibody measurements (IgA + IgG) and pathogen detection (multiplex PCR). Simultaneous measurement of multiple biomarkers allows the analysis of interactions between innate and adaptive immune immunity and pathogen density at the mucosal level. The total number of children will be divided into discovery and validation cohorts. The discovery cohort included an age- and sex-balanced cohort of 80 children: 40 with a severe course and 40 with relatively mild infection (80/80 already included). The results from all markers are used to create a classification model that selects a limited number of markers that are then tested in the here proposed second independent validation cohort of a minimum of 236 children with an acute RTI (see power calculation below). Markers with a persistently high discriminatory value in the validation cohort will be compared for performance against standard clinical diagnostic measurements in serum (including CRP) for their performance in assessing severity and the potential need for antibiotic treatment.

Initial data from analysed work allows for the following power calculation:

Power calculation: For the discovery cohorts, 40 children per group is needed to achieve 80% power for each of n=100 tests (individual test alpha = 0.00090) to detect an actual mean difference of 0.6 with expected SD per group 0.6, applying a false discovery rate (FDR) of 0.010 using a two-sided Mann-Whitney U test.10,11 For the inclusion of the here proposed validation cohort, there is an anticipated 25% severe infections and an alternative AUC of 0.85 - 0.90. Conservatively taking an AUC of 0.77 under the alternative hypothesis, a sample of 59 is needed from the severe group and 138 from the mild group to reject the same null hypothesis AUC of 0.65 with 80% power. Thus, there is a need to include a minimum total of (100/25*59) = 236 children in the acute RTI validation cohort. By anticipating a 10% dropout rate, the minimum total number of children that is aimed to include is 260 (up to 300 inclusions in the case of a higher-than-expected dropout rate).

IBM SPSS Statistics software (SPSS Statistics for Windows; IBM, Armonk, NY) and or STATA will be used for analysis. Demographic and clinical characteristics will be described using standard statistical analysis methods. The descriptive data will be presented as percentages and medians ± interquartile range, or numbers with percentages.Ethical considerations The study will be conducted according to South African and internationally accepted ethical standards, including the Declaration of Helsinki and the South African Good Clinical Practice Guidelines (SA GCP). An annual progress report with intermediate results will be submitted to the Ethics committee and funders. In addition, records will be available to HREC for inspection (quality assurance and compliance with regulations), while always maintaining participant confidentiality.

Informed consent and assent Parents/ legal guardians, or in special cases caregivers, of the child, will be required to give informed consent for the child's participation in the study. Legal guardians will be required to produce documentation to prove legitimate guardianship. In some cases, we will allow a primary caregiver to give informed consent. This will be considered when there are no parents or legal guardians around and the caregiver has a clear history of being the primary caregiver of the child. In addition, this exception will be discussed with the HREC committee. Oral and written information about the study and study procedures will be given, together with the consent form in the preferred language (English, Afrikaans, isiXhosa). An interpreter will be used if necessary. Children > 7 years of age will also have to sign assent for the study. The child/ parent/legal guardian/ caregiver will be able to withdraw the child from the study at any time point, without this adversely affecting the standard care.

A copy of the signed Informed Consent/Assent Form along with a copy of the most recent approved Patient Information Sheet will be given to the study participant. An original signed and dated consent form will be retained in the Investigator Site File (ISF) and a copy will be placed in the medical notes. This consent, and ethical approval, covers the future laboratory analysis of blood and respiratory samples taken during this study.

Privacy and confidentiality The identity of all study subjects will be protected by adhering to all SA GCP guidelines on data handling and storage.

Storage of paper data During the data collection phase, paper-based data will be stored in fire-resistant locked cabinets in a dedicated, locked room. They will be transported in locked bags/boxes to and from research sites/rooms.

After data collection has been completed and the database is clean and locked for analysis, all paper-based data will be securely archived either offsite with a company that specializes in archival, or onsite in a dedicated storage space in fire-resistant cabinets. This will be for the duration required by SA GCP. The longest required timeline will be taken as the archival time. Once this time is completed, the PI will be asked to authorize the destruction of all paper-based forms.

Data-management At recruitment, each patient will be assigned a unique anonymous study barcode. All documents and samples related to a single participant will be marked with the participant's unique barcode. No identifying data will appear on the samples. Only the consent form and demographic form (containing the subject's contact details necessary for follow-up tracing) will have the subject's personal information linked to the barcode- these documents will be stored separately from the other documents in a locked cabinet at DTTC. Samples will be stored in dedicated freezers at the DTTC, where technical and maintenance support is available on a 24-hour basis. All data will be stored without personal identifiers; lab personnel will be blinded to clinical and personal data. Data will be stored on protected servers at DTTC with limited access by the database manager, PI and selected co-investigators only. No other genetic testing will be performed unless permission is requested and granted from the HREC.

Potential harm/ risk Overall, the procedures in this proposed work have minimal risk to study participants. Routine care procedures are carried out by qualified health care professionals according to the Health Professions Council of South Africa (HPCSA).

Routine care data and sample collection All procedures (CXR, HIV testing and respiratory sample collection) are standard of care and are routinely recommended and performed in the study setting to investigate children with respiratory illness, with limited patient risk.

Respiratory sampling: NPAs or NPSs cause mild discomfort and a minimal risk of nosebleeds. After instilling a few drops of sterile saline solution into both nostrils, mucus is aspirated from the posterior nasopharynx using a soft cannula attached to a mucus extractor. The procedure lasts a couple of minutes.

For NPA collection, the suction machine is set at a pressure that will not cause major trauma to the mucosal lining of the nose and throat. Suction pressures by age, according to the American Association for Respiratory Care (AARC) Guidelines for appropriate sub-atmospheric nasotracheal suctioning pressures, will be followed:

Neonates: 60 - 80 mm Hg (0.079- 0.10 Bar) Infants: 80 - 100 mm Hg (0.079- 0.13 Bar) Children: 100 - 120 mm Hg (0.13- 0.15 Bar)

All procedures of this proposed research are minimally invasive with very limited risk for the participants. The study personnel will be committed to minimising risks to the child at all times. The study nurse will be trained in all study investigations and will follow strict standard operating procedures with the help of a research assistant.

The collection of NPAs will take place in a well-ventilated room, and particulate N95 respirators and goggles or protective eye screens will be worn throughout the procedure to protect parents and healthcare providers from possible respiratory pathogen (including TB) aerosolization.

Radiology: Chest radiographs (CXR) will only be taken at enrolment if clinically indicated. The total radiation dose per child is approximately 0.05 mSv (depending on age and including antero-posterior and lateral films), which is roughly equivalent to 30 days of background environmental exposure (Duke University Radiation Safety Committee, IRB Protocol Radiation Risk Statements. Website: http://www.safety.duke.edu/RadSafety).

Phlebotomy: Children may experience pain associated with phlebotomy. A maximum of three attempts will be made to obtain the venous blood specimen. Arterial blood specimens will not be obtained. The study nurse and physician will be experienced and trained to perform phlebotomy. Additionally, local analgesia and distracters such as toys and music will be used to minimize stress experienced by children.

The HREC guideline for the SOP for researchers will be used when determining what volume of blood can be used for research purposes. Internationally accepted and NIH research guidelines regarding study involvement of children dictate that children should provide no more than 3% of total blood volume per 24-hour period (www.irb.pitt.edu/Guidance/Bloodwithdrawpediatrics.pdf). Thus, venous blood specimens provided by study participants are generally considerably less than the recommended guidelines. For children weighing less than 5kg, the blood draw for serum will be restricted to 1.5ml. This will still enable sufficient serum for the primary aim of the study, but there will be less for storage for planned future work. To minimize risk and in consideration of culturally accepted norms, we will exclude children who weigh < 2.5 kg. Ill children who are on intravenous rehydration infusions or anaemic (Hb<8.5), will have the initial procedures deferred.

Cost to parent/legal guardian All study procedures will be paid for from study funds i.e. there will be no cost to the study participant or their family. The parent/legal guardian will receive a small payment for participation in the study (time and inconvenience) while seen in hospital. The South African Health Product Regulatory Authority Clinical Trial Participant Time, Inconvenience and Expense (TIE) Compensation Model will be adhered to, and the enrolment will likely last <3 hours and consequently reimbursement for time will be ± 150 ZAR for enrolment. The enrolment and sampling will occur at TBH during hospital admission only. Child and caregiver are not expected to come back.

Infection control measures Safe handling of bio-hazardous material All team members involved in obtaining biological specimens will be trained in the safe handling of such materials. Sharps used for blood taking will be disposed of safely and rapidly into a dedicated sharps container.

All laboratory facilities linked to the proposed work are well-established and accredited to work with bio-hazardous materials.

Protection from potentially infectious respiratory secretions All team members involved in obtaining NPAs from study participants will wear N95 respirator masks, which will be fit tested once yearly on all staff. The procedures will be undertaken in a dedicated sampling room with an extraction fan and according to DTTC infection control SOP.

ELIGIBILITY:
Inclusion Criteria:

- Children aged 0-13 years with acute respiratory tract infections presenting to Tygerberg Hospital (TBH) in Cape Town, South Africa, for routine care

Exclusion Criteria:

* Admitted for < 72 hours

Max Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 0-13 years will be recruited from Tygerberg Hospital (TBH) in Cape Town, South Africa. TBH serves as regional referral centres to the surrounding health sub-districts (Northern, Tygerberg, Khayelitsha and Eastern) serving over 30% of the metropolitan population (3.5 million residents). TBH also serves as a tertiary-level referral centre for paediatric emergencies, infectious diseases and pulmonology.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-10-23 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Poly-reactive and pathogen-specific antibodies in the saliva and serum of South African children presenting with an acute respiratory tract infection to Tygerberg Hospital. | Antibodies will be measured at baseline (enrolment) in saliva and serum and in saliva on the second and third day of admission and on the day of discharge (up to 90 days from baseline).
  Total antibodies to specific respiratory pathogens, as well as poly-reactive antibodies (IgG, IgA and IgM), will be measured in serum and saliva at the time of presentation to hospital. In addition, antibodies will be measured in saliva on days 2 and 3 of admission and on the day of discharge up to 90 days from baseline. The percentage of polyreactive antibodies to pathogen-specific antibodies will be calculated.
Targeted protein markers in the saliva and serum of children presenting to Tygerberg Hospital with an acute respiratory tract infection. | Inflammatory protein markers will be measured in saliva and serum at baseline, with additional saliva measurements on days 2 and 3 of admission and on the day of discharge (up to 90 days).
  Protein markers in saliva and serum will be measured using a Luminex based Multiplex Immuno-Assay (MIA). Inflammatory markers that will be measured include: CCL19, CCL20, CCL28, CXCL11, CCL11, HGF, CXCL5, CXCL6, IFN-y, TNF-a, MMP2, MPO, Procalcitonin, CRP, and IL-6. All markers will be measured in ug/ml.
The respiratory pathogens identified in children presenting to Tygerberg Hospital with acute respiratory illnesses | Nasopharyngeal aspirates will be done at baseline (day of enrolment).
  Nasopharyngeal aspirates will be done on all children at enrolment. The Allplex™ RV Essential Assay and a COVID PCR will be done on the NPA samples. The RV 7 tests for 7 viruses: Adenovirus (AdV), Influenza A virus (Flu A), Influenza B virus (Flu B), Metapneumovirus (MPV), Parainfluenza virus (PIV), Respiratory syncytial virus (RSV), Human rhinovirus A/B/C (HRV).

SECONDARY OUTCOMES:
Severity of respiratory disease in South African children presenting with acute respiratory tract infections to Tygerberg Hospital. | Severity of respiratory distress will be quantified at baseline (presentation to hospital) and at discharge (up to 90 days from baseline).
  Severity of disease will be determined at presentation and discharge according to the Clinical Respiratory Distress (CRS) score. The CRS uses 6 parameters to obtain a score. These include respiratory rate, auscultation, use of accessory muscles, mental status, room air saturations and colour. Respiratory distress is then classified into mild, moderate or severe. 0-3: Mild distress; 4-6: Moderate distress; ≥7: Severe distress.
  Data will be captured on CRFs from the time of admission to the time of hospital discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Marieke van der Zalm, PhD, Principal Investigator — Desmond Tutu TB Centre
Locations (2):
- South Africa (2):
  - Desmond Tutu TB Centre, Tygerberg Hospital, Cape Town, Western Cape
  - Desmond Tutu TB Centre, Cape Town, Western Cape

IPD SHARING:
Plan to Share IPD: Undecided
This will depend on local ethics review board advice and discussion with community advisory board.

REFERENCES:
- [Background] Anthony MG, Hoddinott G, Van Niekerk M, Dewandel I, McKenzie C, Bekker C, Rabie H, Redfern A, van der Zalm MM. The socioeconomic impact of the COVID-19 lockdown on families affected by childhood respiratory illnesses in Cape Town, South Africa. PLOS Glob Public Health. 2024 Mar 28;4(3):e0003020. doi: 10.1371/journal.pgph.0003020. eCollection 2024. PMID 38547177
- [Background] Bekker C, Dewandel I, Redfern A, McKenzie C, Lishman J, Verhagen LM, Claassen M, Wilson S, Dunbar R, Bosch C, van Zyl G, Preiser W, Goussard P, Rabie H, van der Zalm MM. Clinical spectrum of disease and outcomes in children with Omicron SARS-COV-2 infection in Cape Town, South Africa. IJTLD Open. 2024 Jan 1;1(1):27-33. doi: 10.5588/ijtldopen.23.0053. eCollection 2024 Jan. PMID 38919411
- See also: VERDI is a project that prioritises pregnant women, children and high-risk populations in research on new SARS-CoV-2 variants of concern. It also focuses on preparedness for future infections outbreaks, building on experiences with COVID-19 and mpox. — https://verdiproject.org/